CLINICAL TRIAL: NCT04602234
Title: Diagnosis of Lower Respiratory Tract Infection by Lung Ultrasonography in General Practice : a Prospective, Interventional and Multicentric Study
Brief Title: Diagnostic of Lower Respiratory Tract Infection by Lung Ultrasonography in General Practice
Acronym: AmbuLUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-A00205)52
Record Dates: First submitted 2020-10-20; First posted 2020-10-26 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Lower Resp Tract Infection; Ultrasound Therapy; Complications
Keywords: Lung ultrasonography; Lower Respiratory Tract Infection; General Practice

STUDY DESIGN:
Intervention Model Description: Among the 151 patients included, 111 LUS were performed (LUS group)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LUS group (Experimental)
  Interventions: Diagnostic Test: Lung ultrasonography
- No LUS group (No Intervention)

INTERVENTIONS:
Diagnostic Test: Lung ultrasonography — Investigators performed lung ultrasonography on patients
  Arms: LUS group

SUMMARY:
Lower Respiratory Tract Infection (LRTI) is a frequent motive of consultation in General Practice. Cost, irradiation and availability of traditional imagery make it difficult to perform in every patient with suspected LRTI.

The objective is to evaluate the performance of LUS realized by family physicians into the usual LRTI diagnostic pathway.

This study is a prospective, interventional, multi-centric and open study conducted in 3 different centers by 15 General Practitioners (GP) in France. Patient complaining of dyspnea or cough were recruited from December 2019 to March 2020. GP received a training course by LUS expert before the study.

The primary outcome measure was diagnosis modification after LUS. Secondary measures were therapeutic modification after LUS, decision of imagery prescription after LUS, decision of hospitalization or not after LUS, medical evolution and result of imagery initially prescribed by GP.

DETAILED DESCRIPTION:
After an initial medical report, GP's concluded to an initial diagnosis and make initial prescription and finally decided or not to perform a standardized eight-points LUS. GP were free to perform or not LUS. If GP decided to perform LUS, GP were allowed to change their diagnosis and prescriptions (LUS group). However, therapeutic changes after LUS could not "downgrade" patient care.

ELIGIBILITY:
Inclusion Criteria:

* Age > 3 months
* Dyspnea or cough complaint

Exclusion Criteria:

* Age < 3 months
* Rejection to participate to the study

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2019-12-30 (Actual); Primary Completion 2020-03-11 (Actual); Study Completion 2020-03-18 (Actual)

PRIMARY OUTCOMES:
Diagnosis modification | 3 months
  Diagnosis modification after lung ultrasonography

SECONDARY OUTCOMES:
Therapeutic modification | 3 months
  Therapeutic modification after lung ultrasonography
Imagery prescription | 3 months
  Decision of imagery prescription after lung ultrasonography
Decision of hospitalization | 3 months
  Decision of an hospitalization or not after lung ultrasonography
Medical evolution | 3 months
  Medical evolution at 7 days (improvement, persistence, worsening and hospitalization)
Imagery result | 3 months
  Result of imagery initially prescribed by general practitioners (Chest CT-Scan or X-Ray)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Caen, Caen, Calvados, France

REFERENCES:
- [Derived] Amiot F, Delomas T, Laborne FX, Ecolivet T, Macrez R, Benhamed A. Implementation of lung ultrasonography by general practitioners for lower respiratory tract infections: a feasibility study. Scand J Prim Health Care. 2024 Sep;42(3):463-470. doi: 10.1080/02813432.2024.2343678. Epub 2024 May 20. PMID 38767949